CLINICAL TRIAL: NCT06865755
Title: Deploying and Evaluating a Technology Based System to Help People Adhere to Long Term Medications
Brief Title: Collaborative Research: Multiscale Modeling and Intervention for Improving Long-Term Medication
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: University of Virginia (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kristen Wells, Professor, San Diego State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HS-2024-0145; R01CA239246 (NIH)
Record Dates: First submitted 2024-10-15; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer Survivor; Breast Cancer Early Stage Breast Cancer (Stage 1-3)
Keywords: Single-Arm Study Design; Medication Event Monitoring System (MEMS); Medication Adherence; Breast Cancer Survivors; Personalized Interventions; endocrine therapy; mobile health
MeSH Terms: conditions — Medication Adherence | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- integrated medication monitoring system (Experimental): The single-arm intervention design of this study focuses on delivering a comprehensive integrated medication monitoring system to a cohort of breast cancer survivors. The system will analyze data collected from EMAs, MEMS, and Fitbit sensors to identify participants at risk of nonadherence. Based on this risk assessment, personalized interventions will be delivered through the Digital Trails app, which may include reminders for medication intake, among others.
  Interventions: Device: integrated medication monitoring (MM) system

INTERVENTIONS:
Device: integrated medication monitoring (MM) system — We have created a new integrated medication monitoring (MM) system consisting of baseline, 3-month, and 6-month surveys, smartphone-based ecological momentary assessment via an application installed on a smartphone (Digital Trails based on the UVA Sensus app), a wireless medication event monitoring system device (MEMS; Wisepill), and a wearable sensor (Fitbit), and data collected passively from smartphone sensors using the Digital Trails app. These sources of information will be used to understand predictors of medication taking behaviors and, after two months of monitoring, to deploy appropriate interventions which will be delivered via the Digital Trails app platform.

SUMMARY:
The goal of this study is to learn about the impact of an integrated medication monitoring system in breast cancer survivors aged 21-70 who are prescribed endocrine therapy. The main question it aims to address is: Does the integrated medication monitoring system improve medication adherence among breast cancer survivors when used over a six-month period?

Fifteen English-speaking breast cancer survivors who meet the inclusion criteria will use a combination of smartphone-based ecological momentary assessments, a medication event monitoring system (Wisepill), and a wearable sensor (Fitbit). After 2 months, participants will be provided personalized content to facilitate medication adherence through an app (Digital Trails) and through WisePill. Participants will complete online surveys at baseline, 3 months, and 6 months to assess their experiences and adherence.

DETAILED DESCRIPTION:
Purpose/objective:

The investigators have created a new integrated medication monitoring (MM) system for long-term monitoring of medication adherence consisting of baseline, 3-month, and 6-month surveys, smartphone based ecological momentary assessment, smartphone sensors, a medication event monitoring system (MEMS; Wisepill) sensor, and a wrist-worn wearable sensor (Fitbit) that will be used to collect data to understand and model medication-taking behaviors. The objective of the project is to deploy this system to predict nonadherence to endocrine therapy for breast cancer survivors and implement intervention strategies to improve medication adherence. These interventions will be evaluated for preliminary impact on behavior, acceptability, attractiveness, and usefulness.

Overview:

The investigators will conduct a single arm study collecting data in multiple ways and multiple intervals, over six months' time: 1) baseline, 3-month, and 6-month surveys via Qualtrics; 2) smartphone-based ecological momentary assessment (via Digital Trails application) at the following intervals: every 2-3 days, weekly, and monthly; 3) wireless medication event monitoring system devices (MEMS; Wisepill; daily), 4) a wrist-worn wearable sensor (Fitbit; continuous); and 5) smartphone sensors (data collected via Digital Trails application, continuous). Participants will be provided personalized intervention content based on their specific risk via the Digital Trials app. Fifteen breast cancer survivors will be asked to participate in this longitudinal study for six months.

Intervention:

The investigators have created a new integrated medication monitoring (MM) system consisting of baseline, 3-month, and 6-month surveys, smartphone-based ecological momentary assessment via an application installed on a smartphone (Digital Trails based on the UVA Sensus app), a wireless medication event monitoring system device (MEMS; Wisepill), and a wearable sensor (Fitbit), and data collected passively from smartphone sensors using the Digital Trails app. These sources of information will be used to understand predictors of medication taking behaviors and, after two months of monitoring, to deploy appropriate interventions which will be delivered via the Digital Trails app platform. The objective of the project is to deploy this MM system to predict nonadherence to endocrine therapy for breast cancer survivors and implement intervention strategies to improve medication adherence (via Digital Trails). These interventions will be evaluated for preliminary impact on behavior, acceptability, attractiveness, and usefulness.

Participant Eligibility Criteria Fifteen breast cancer survivors will be included in the study if they: 1) are English-speaking and reading; 2) are between ages 21 and 70 years; 3) are diagnosed with stage 0-3 breast cancer in the past 5 years; 4) have completed all surgery, radiation, and chemotherapy, except endocrine therapy; 5) are prescribed endocrine therapy; 6) do not have a physical impairment that would prevent them from using the MM system; 7) are able to provide informed consent; 8) are willing and able to use the MM system for 6 months; and 9) have an Iphone or Android phone.

Participant Recruitment Using convenience sampling, the investigators will recruit 15 breast cancer survivors. The study will be publicized using a number of different ways, including ads on social media. Participants will be directed to complete an online screening survey via Qualtrics or to contact the study staff via email or phone. The investigators will contact interested participants and do a telephone or HIPAA-Zoom screening to assess study inclusion criteria, after obtaining informed consent. The investigators will then provide sensors to participants (via mail) and in a subsequent baseline data collection session (via Zoom), assist participants with completing baseline surveys via Qualtrics, in learning how to use the sensors, and in downloading and using smartphone applications. Participants will be asked to use two sensors: 1) a medication event monitoring system device (MEMS; Wisepill); and 2) a wrist-worn wearable sensor (Fitbit) daily for the next 6 months (see below). Participants will be asked to download the Fitbit and Digital Trails apps to their smartphones. Participants will also be asked to complete ecological momentary assessment (EMA; short surveys) using a smartphone app (Digital Trails) for six months.

Data Collection Digital Trails is an app that combines Sensus, a novel mobile sensing system for Android and iOS capable of collecting data from smartphone and Bluetooth-enabled sensors and administering EMAs, with a smartphone intervention. EMA surveys will be implemented at the following intervals: 1) randomly; 2) every 2- 3 days; 3) every 14 days; and 4) every 28 days. Digital Trails will also collect data from the participants' smartphone if authorized by the participant. These may include, but are not limited to, GPS, accelerometer, gyroscope, and pedometer data. Participants will complete 3 surveys via Qualtrics, at baseline, three month follow-up, and six-month follow-up. These surveys will be administered via Qualtrics. Participants will be asked to use two sensors daily for the entire six month period: 1) a Fitbit wrist sensor; and 2) a Wisepill MEMS cap. The investigators will use the Fitbit Sense smartwatch to collect data including steps, calories burned, total distance traveled, sleep, flights of stairs climbed, active minutes, exercise, and average heart rate. Participants will be asked to download the Fitbit app onto their personal smartphone. Participants' Fitabase data will be monitored by the study team using the Fitabase dashboard.

Primary Outcomes: Adherence to medication, receipt of intervention components, perception of intervention (thoughts, most useful components, lease useful components, most attractive components, least attractive components, problems with the intervention, suggested changes to intervention, additional information that should be provided by intervention, willingness to use intervention/system in future).

Planned analyses:

Evaluation of immediate response to delivery of each intervention module will consist of examining MM data that measure: 1) detection of a risk for missed medication; 2) delivery of the specific intervention module suggested by our modeling; and 3) whether the participant subsequently took the medicine as prescribed after the intervention module was deployed (within a 24 hour interval from the last dose plus or minus 6 hours). The investigators will also summarize data regarding participants' use of each type of module offered and their assessment of the acceptability, attractiveness, and usefulness of intervention modules used. Data collected from close-ended questions (i.e., use of an intervention module) will be summarized using descriptive data (i.e., counts and frequencies). Qualitative data collected from open-ended questions will be summarized using content analysis by having two raters code data on the three a priori themes (i.e., acceptability, attractiveness, and usefulness).

ELIGIBILITY:
Inclusion Criteria:

* are English-speaking and reading;
* are between ages 21 and 70 years;
* are diagnosed with stage 0-3 breast cancer in the past 5 years;
* have completed all surgery, radiation, and chemotherapy, except endocrine therapy;
* are prescribed endocrine therapy;
* do not have a physical impairment that would prevent them from using the MM system;
* are able to provide informed consent;
* are willing and able to use the MM system for 6 months;
* have an Iphone or Android phone.

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Wisepill MEMS Sensor data collection | From enrollment to the end of study at 6 months
  Participants will be asked to put their endocrine therapy medication in the Wisepill device and will be asked to open the Wisepill when taking their medicine daily for six months
Intervention component - Introduction | 6 months after enrollment into study
  Number of respondents who reported receiving and/or using the app introduction
Intervention component - Instructions | 6 months after enrollment into the study
  Number of respondents who reported receiving and/or using instructions for using the app
Intervention component - calendar | 6 months after enrollment into the study
  Number of respondents who reported receiving and/or using the app calendar
Intervention component - resources | 6 months after enrollment into the study
  Number of respondents who reported receiving and/or using resources for breast cancer survivors
Intervention component - relaxation audio files | 6 months after enrollment into the study
  Number of respondents who reported receiving and/or using relaxation audio files
Intervention component - social support | 6 months after enrollment into the study
  Number of respondents who reported receiving and/or using information about social support
Intervention component - tamoxifen | 6 months after enrollment into the study
  Number of respondents who reported receiving and/or using information about tamoxifen
Intervention component - aromatase inhibitors | 6 months after enrollment into the study
  Number of respondents who reported receiving and/or using information about aromatase inhibitors
Intervention component - routine | 6 months after enrollment into the study
  Number of respondents who reported receiving and/or using information about establishing a routine for taking medications
Intervention component - reminders | 6 months after enrollment into the study
  Number of respondents who reported receiving and/or using information about setting medication reminders
Intervention component - joint pain | 6 months after enrollment into the study
  Number of respondents who reported receiving and/or using information about managing joint pain
Intervention component - hot flashes | 6 months after enrollment into the study
  Number of respondents who reported receiving and/or using information about managing hot flashes
Intervention component - pacing | 6 months after enrollment into the study
  Number of respondents who reported receiving and/or using information about pacing
Intervention component - relaxation | 6 months after enrollment into the study
  Number of respondents who reported receiving and/or using information about relaxation
Intervention component - needs | 6 months after enrollment into the study
  Number of respondents who reported receiving and/or using information about getting what they need from their health care providers
Intervention component - travel | 6 months after enrollment into the study
  Number of respondents who reported receiving and/or using information about travel
Intervention component - thoughts | 6 months after enrollment into the study
  Participants will be asked to describe what they thought about the intervention overall (qualitative response)
Intervention component - most useful | 6 months after enrollment into the study
  Participants will be asked to describe the most useful intervention components (qualitative response)
Intervention component - least useful | 6 months after enrollment into the study
  Participants will be asked to describe the least useful intervention components (qualitative response)
Intervention component - most attractive | 6 months after enrollment into the study
  Participants will be asked to describe which intervention components were most attractive (qualitative response)
Intervention component - least attractive | 6 months after enrollment into the study
  Participants will be asked to describe which intervention components were least attractive (qualitative response)
Intervention component - problems | 6 months after enrollment into the study
  Participants will be asked to describe problems they experienced using the intervention application (qualitative response)
Intervention component - changes | 6 months after enrollment into the study
  Participants will be asked to describe any changes they would make to the intervention (qualitative response)
Intervention component - additional information | 6 months after enrollment into the study
  Participants will be asked to describe what additional information the intervention should provide (qualitative response)
Intervention component - future use | 6 months after enrollment into the study
  Participants will be asked to describe whether or not they would be willing to use the intervention and monitoring system in the future to remember to take medicines.

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share the data so it can be anonymized in registries such as Open Science Framework or alongside our publications.